CLINICAL TRIAL: NCT06437197
Title: Clinical and Radiographic Evaluation of Platelets Rich Fibrin in Adult Pulpotomy: Randomized Clinical Trial
Brief Title: Evaluation of Using Platelet-Rich Fibrin in Adult Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Ahmed Qandeel, Demonstrator of Endodontics, Faculty of Dental Medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 867/2992
Record Dates: First submitted 2023-02-09; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy; Platelet Rich Fibrin
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydraulic Calcium Silicate Cement (Active Comparator): Pulpotomy of adult teeth using Hydraulic Calcium Silicate Cement.
  Interventions: Procedure: Pulpotomy
- platelet rich fibrin (PRF) (Experimental): Pulpotomy of adult teeth using platelet Rich fibrin.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — Removal of the coronal pulp chamber in an adult teeth
  Other Names: Pulp amputation

SUMMARY:
The goal of this interventional randomized clinical trial is to evaluate the use of platelet rich fibrin in full pulpotomy in mature adult teeth.

The main questions it aims to answer are:

1. Does the use of platelet rich fibrin in complete pulpotomy in mature permanent teeth will raise the success rate of full pulpotomy of adult teeth?
2. Does the use of cone beam computed tomography scans will be more effective in early detection of apical periodontitis than periapical radiographs?

Participants will be asked to do the following:

* Receive the pulpotomy treatment of their target tooth.
* Record the pain score in the pain assessment chart.
* Attend the follow-up visits. They'll receive a full pulpotomy treatment of their target tooth. Researchers will evaluate the usage of platelet rich fibrin in performing the pulpotomy procedure of adult teeth and if cone beam computed tomography scans will be more effective in early detection of apical periodontitis than periapical radiographs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age: 25-35 years
2. Mature permanent premolar teeth with two separate roots.
3. Clinical diagnosis of irreversible pulpitis.
4. Patients without existing medical condition.

Exclusion criteria:

1. Immature teeth.
2. Non-restorable teeth.
3. Non-vital Teeth.
4. Uncontrolled pulpal bleeding.
5. Periodontally affected teeth.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Radiographic changes in periapical area using periapical radiographs. | 6 and 12 months.
  The radiographic changes was evaluated using periapical radiographs. the outcome was measured using the periapical index scoring 1,2,3,4 or 5 with 1 indicating normal and 5 indicates severe periodontitis with exacerbating features.

SECONDARY OUTCOMES:
Postoperative pain | Immediately, 24, 48, 72 hours and 7 days.
  The postoperative pain was measured by modified modified Visual analog scale VAS which is is segmented into ten levels according to severity of pain, no pain (0), mild pain (1-3), moderate pain (4-6), or severe pain (7-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaculli F, Rodriguez-Lozano FJ, Briseno-Marroquin B, Wolf TG, Spagnuolo G, Rengo S. Vital Pulp Therapy of Permanent Teeth with Reversible or Irreversible Pulpitis: An Overview of the Literature. J Clin Med. 2022 Jul 11;11(14):4016. doi: 10.3390/jcm11144016. PMID 35887779
- [Background] Hanna SN, Perez Alfayate R, Prichard J. Vital Pulp Therapy an Insight Over the Available Literature and Future Expectations. Eur Endod J. 2020 Mar 1;5(1):46-53. doi: 10.14744/eej.2019.44154. eCollection 2020. PMID 32342038
- [Background] Guideline on Pulp Therapy for Primary and Immature Permanent Teeth. Pediatr Dent. 2016 Oct;38(6):280-288. No abstract available. PMID 27931467
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Background] Cervino G, Laino L, D'Amico C, Russo D, Nucci L, Amoroso G, Gorassini F, Tepedino M, Terranova A, Gambino D, Mastroieni R, Tozum MD, Fiorillo L. Mineral Trioxide Aggregate Applications in Endodontics: A Review. Eur J Dent. 2020 Oct;14(4):683-691. doi: 10.1055/s-0040-1713073. Epub 2020 Jul 29. PMID 32726858
- [Background] Cushley S, Duncan HF, Lappin MJ, Tomson PL, Lundy FT, Cooper P, Clarke M, El Karim IA. Pulpotomy for mature carious teeth with symptoms of irreversible pulpitis: A systematic review. J Dent. 2019 Sep;88:103158. doi: 10.1016/j.jdent.2019.06.005. Epub 2019 Jun 20. PMID 31229496
- [Background] Linsuwanont P, Wimonsutthikul K, Pothimoke U, Santiwong B. Treatment Outcomes of Mineral Trioxide Aggregate Pulpotomy in Vital Permanent Teeth with Carious Pulp Exposure: The Retrospective Study. J Endod. 2017 Feb;43(2):225-230. doi: 10.1016/j.joen.2016.10.027. Epub 2016 Dec 29. PMID 28041685
- [Background] Qudeimat MA, Alyahya A, Hasan AA. Mineral trioxide aggregate pulpotomy for permanent molars with clinical signs indicative of irreversible pulpitis: a preliminary study. Int Endod J. 2017 Feb;50(2):126-134. doi: 10.1111/iej.12614. Epub 2016 Feb 22. PMID 26841969
- [Background] Taha NA, Khazali MA. Partial Pulpotomy in Mature Permanent Teeth with Clinical Signs Indicative of Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2017 Sep;43(9):1417-1421. doi: 10.1016/j.joen.2017.03.033. Epub 2017 Jun 30. PMID 28673494
- [Background] Awawdeh L, Al-Qudah A, Hamouri H, Chakra RJ. Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine: A Prospective Randomized Clinical Trial. J Endod. 2018 Nov;44(11):1603-1609. doi: 10.1016/j.joen.2018.08.004. Epub 2018 Oct 3. PMID 30292451
- [Background] Asgary S, Eghbal MJ, Shahravan A, Saberi E, Baghban AA, Parhizkar A. Outcomes of root canal therapy or full pulpotomy using two endodontic biomaterials in mature permanent teeth: a randomized controlled trial. Clin Oral Investig. 2022 Mar;26(3):3287-3297. doi: 10.1007/s00784-021-04310-y. Epub 2021 Dec 2. PMID 34854987
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Borie E, Olivi DG, Orsi IA, Garlet K, Weber B, Beltran V, Fuentes R. Platelet-rich fibrin application in dentistry: a literature review. Int J Clin Exp Med. 2015 May 15;8(5):7922-9. eCollection 2015. PMID 26221349
- [Background] Patidar S, Kalra N, Khatri A, Tyagi R. Clinical and radiographic comparison of platelet-rich fibrin and mineral trioxide aggregate as pulpotomy agents in primary molars. J Indian Soc Pedod Prev Dent. 2017 Oct-Dec;35(4):367-373. doi: 10.4103/JISPPD.JISPPD_178_17. PMID 28914251
- [Background] Eid A, Mancino D, Rekab MS, Haikel Y, Kharouf N. Effectiveness of Three Agents in Pulpotomy Treatment of Permanent Molars with Incomplete Root Development: A Randomized Controlled Trial. Healthcare (Basel). 2022 Feb 25;10(3):431. doi: 10.3390/healthcare10030431. PMID 35326909
- [Background] Keswani D, Pandey RK, Ansari A, Gupta S. Comparative evaluation of platelet-rich fibrin and mineral trioxide aggregate as pulpotomy agents in permanent teeth with incomplete root development: a randomized controlled trial. J Endod. 2014 May;40(5):599-605. doi: 10.1016/j.joen.2014.01.009. Epub 2014 Mar 6. PMID 24767550
- [Background] Noor Mohamed R, Basha S, Al-Thomali Y. Efficacy of platelet concentrates in pulpotomy - a systematic review. Platelets. 2018 Jul;29(5):440-445. doi: 10.1080/09537104.2018.1445844. Epub 2018 Mar 14. PMID 29537945
- [Background] Kumar V, Juneja R, Duhan J, Sangwan P, Tewari S. Comparative evaluation of platelet-rich fibrin, mineral trioxide aggregate, and calcium hydroxide as pulpotomy agents in permanent molars with irreversible pulpitis: A randomized controlled trial. Contemp Clin Dent. 2016 Oct-Dec;7(4):512-518. doi: 10.4103/0976-237X.194107. PMID 27994420
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221